CLINICAL TRIAL: NCT00000449
Title: Coping, Exposure, and Naltrexone Treatment With Alcoholics
Brief Title: Behavior and Naltrexone Treatment for Alcoholics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Factorial | Purpose: Treatment
Other Study IDs: NIAAAMON7850
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: naltrexone (Revia)
Behavioral: cognitive behavioral therapy
Behavioral: cue exposure treatment

SUMMARY:
The study's purpose is to improve alcoholism treatment by investigating the combined effectiveness of a psychotherapy (Coping Skills Training and Cue Exposure Treatment - CSTCET) with naltrexone in a randomized clinical trial. Individuals will receive 2 weeks of CSTCET or a control treatment as inpatients followed by 12 consecutive weeks of receiving either naltrexone or placebo as outpatients. Followups at 24, 48, and 72 weeks after treatment is completed.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence.

Exclusion Criteria:

* Current diagnosis of dependence on other substances except nicotine.
* A history of psychosis or current psychotic symptoms.
* Current suicidality, homocidality, or psychiatric symptoms that require additional medication.
* Current use of disulfiram (Antabuse).
* Evidence of significant cerebral, renal, thyroid, or cardiac disease.
* History of opioid abuse in the previous year.
* History of cirrhosis, hepatocellular disease, or elevated bilirubin.
* Females who are pregnant, nursing, or not using a reliable method of birth control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States